CLINICAL TRIAL: NCT03429738
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Ibuprofen and Pseudoephedrine Hydrochloride 200 mg/30 mg Tablets Under Fasting Conditions
Brief Title: Single-Dose Bioavailability Study of Two Formulations of Ibuprofen and Pseudoephedrine Hydrochloride Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Pharma Medica Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PMRI study number 2014-3489
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Pain, Head; Pain, Acute; Pain, Back; Fever
Keywords: Ibuprofen; phase-I-study; pharmacokinetic; combination therapy; bioavailability; bioequivalence; pseudoephedrine hydrochloride
MeSH Terms: conditions — Headache; Acute Pain; Back Pain; Fever | interventions — Ibuprofen; Pseudoephedrine

STUDY DESIGN:
Intervention Model Description: open-label, single-dose, randomized, two-period, two-treatment, twosequence, crossover, comparative bioavailability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Drug (Experimental): Drug: Ibuprofen/Pseudoephedrine HCl 200/30 mg Film-Coated Tablets Temmler Werke GmbH/ Part of Aenova Group, Germany, Intervention: one tablet administered after an overnight fast of at least 10 hours
  Interventions: Drug: Ibuprofen/Pseudoephedrine HCl 200/30 mg Film-Coated Tablets
- Active Comparator (Active Comparator): Active Comparator: RhinAdvil Rhume 200 mg/30 mg Film-Coated Tablets Wyeth Santé Familiale, France, Intervention: one tablet administered after an overnight fast of at least 10 hours
  Interventions: Drug: RhinAdvil Rhume 200 mg/30 mg Film-Coated Tablets

INTERVENTIONS:
Drug: Ibuprofen/Pseudoephedrine HCl 200/30 mg Film-Coated Tablets — Experimental drug
  Other Names: Ibuprofen/Pseudoephedrine/test product
  Arms: Experimental Drug
Drug: RhinAdvil Rhume 200 mg/30 mg Film-Coated Tablets — Active Comparator
  Other Names: RhinAdvil
  Arms: Active Comparator

SUMMARY:
Evaluation of the comparative bioavailability between two oral formulations containing ibuprofen 200 mg and pseudoephedrine 30 mg after a single dose in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
Ibuprofen is one of the most often used non steroidal antiinflammatory drug (NSAR) in the management of mild to moderate pain and inflammation. Combined with the sympathomimetic pseudoephedrine as decongestant it is widely used in colds or fever. The purpose of this phase-I-study was to evaluate the comparative bioavailability between a combination of 200 mg ibuprofen and 30 mg pseudoephedrine film-coated tablets to the reference formulation RhinAdvil Rhume® 200 mg/30 mg (Wyeth Santé Familiale, France).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking, male and female subjects, 18 years of age or older.
2. BMI ≥ 18.5 and 30.0 kg/m2
3. No clinically significant findings in vital signs measurements.
4. No clinically significant abnormal laboratory values.
5. No clinically significant findings in a 12-lead electrocardiogram (ECG).
6. No significant diseases.
7. Willing to use an acceptable, effective method of contraception.
8. Be informed of the nature of the study and give written consent prior to any study procedure.
9. Have no clinically significant findings from a physical examination.

Exclusion Criteria:

1. Known history or presence of any clinically significant medical condition.
2. Known or suspected carcinoma.
3. History or presence of ulcerative colitis, diverticulosis, Crohn's disease, or gastrointestinal ulcer, perforation, or haemorrhage.
4. Known history or presence of auto-immune disorders, gastrointestinal toxicity, or a risk of gastrointestinal bleeding or gastrointestinal tract irritation.
5. Known history or presence of cardiovascular disease, heart failure, tachycardia, hypertension, angina pectoris, hyperthyroidism, psychosis, seizures, risk of urinary retention, diabetes, phaeochromocytoma, closed angle glaucoma, chronic rhinitis, or prostatic enlargement.
6. Known history or presence of angioedema.
7. Known history or presence of galactose or fructose intolerance, sucraseisomaltase insufficiency, Lapp lactase insufficiency, galactosemia, or glucose-galactose malabsorption syndrome.
8. Known history of severe skin reactions (e.g. exfoliative dermatitis, SJS, and TEN).
9. Known history or presence of bronchial asthma or allergic disease resulting in bronchospasm.
10. Presence of hepatic or renal dysfunction.
11. Presence of clinically significant gastrointestinal disease or history of malabsorption within the last year.
12. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
13. History of drug or alcohol addiction requiring treatment.
14. History of gastrointestinal bleeding or perforation when previously taking NSAIDs.
15. Positive test result for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
16. Positive test result for urine drugs of abuse (cannabinoids, opiates, amphetamines, cocaine, phencyclidine, tricyclic antidepressants, barbiturates, methadone and benzodiazepines) or urine cotinine.
17. Difficulty fasting or consuming standard meals.
18. Does not tolerate venipuncture.
19. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
20. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
21. Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
22. Donation or loss of whole blood (including clinical trials):

    * 50 mL and ≤ 499 mL within 30 days prior to drug administration
    * 500 mL within 56 days prior to drug administration.
23. Females who:

    Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to dosing; Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to drug administration; Are pregnant (serum hCG consistent with pregnancy); or Are lactating.
24. Have had a tattoo or body piercing within 30 days prior to drug administration.
25. Known history or presence of hypersensitivity or idiosyncratic reaction to ibuprofen, pseudoephedrine, NSAIDs, or any other drug substances with similar activity or any of the excipients in the drug products
26. Use of drugs in the phenethylamine and amphetamine chemical classes within 14 days prior to drug administration.
27. Use of NSAIDs (including cyclo-oxygenase-2 selective inhibitors) aspirin, corticosteroids, anticoagulants, selective serotonin-reuptake inhibitors, antihypertensives, diuretics, cardiac glycosides, lithium, methotrexate, cyclosporin, mifepristone, tacrolimus, zidovudine, linezolid, dopaminergic alkaloids, quinolone antibiotics, terpene derivatives, clobutinol, atropine, local anaesthetics, MAO inhibitors, vasoconstrictors, alpha sympathomimetic drugs, or anti-platelet agents within 30 days prior to drug administration.
28. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to drug administration. (e.g. barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole, antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-04-27 (Actual); Primary Completion 2014-05-05 (Actual); Study Completion 2014-05-05 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) (area under the analyte concentration versus time curve) of ibuprofen and pseudoephedrine, respectively | 7 days (± 3 hours)
  The 90% confidence intervals of the relative mean plasma (1S,2S)- pseudoephedrine and (S) ibuprofen AUC should be between 80.00 and 125.00%
maximum serum concentration of ibuprofen and pseudoephedrine, respectively | 7 days (± 3 hours)
  The 90% confidence intervals of the relative mean plasma (1S,2S)- pseudoephedrine and (S) ibuprofen Cmax should be between 80.00 and 125.00%

CONTACTS AND LOCATIONS:
Overall Officials: Latifa Yamlahi, MD, Study Director — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
no IPD to be shared